CLINICAL TRIAL: NCT01698177
Title: Optimizing Influenza Vaccination in Surgical Oncology Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 240293
Record Dates: First submitted 2011-08-11; First posted 2012-10-02 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Influenza
Keywords: Influenza; Cancer; Vaccination; Immune response to influenza vaccination
MeSH Terms: conditions — Influenza, Human; Neoplasms | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Active Comparator): This group will receive the influenza vaccine preoperatively.
  Interventions: Biological: Influenza vaccine
- Group B (Active Comparator): Group B will receive the influenza vaccine postoperatively, prior to hospital discharge.
  Interventions: Biological: Influenza vaccine
- Group C (No Intervention): Group C subjects have already received the seasonal flu vaccine.
- Group D (Placebo Comparator): Group D subjects have refused the vaccine, but agree to have serum titers drawn.

INTERVENTIONS:
Biological: Influenza vaccine — Seasonal inactivated trivalent vaccine
  Arms: Group A
Biological: Influenza vaccine — Seasonal inactivated trivalent vaccine
  Arms: Group B

SUMMARY:
Seasonal influenza (flu) is a significant and sometimes serious health issue in the U.S. The Centers for Disease Control (CDC) estimates that over 200,000 people are hospitalized in the U.S each year related to the flu. Public health campaigns advocate widespread vaccination for the flu, and especially for high risk people. People with cancer are high risk, with an increased risk of developing complications from the flu, such as pneumonia, bronchitis, or worsening of other medical conditions. As part of their vaccination campaign, the CDC strongly encourages inpatients to be vaccinated prior to hospital discharge. Accordingly, Stony Brook Hospital has enacted a policy that mandates screening all hospital inpatients for vaccination prior to discharge. While physicians or patients can opt not to vaccinate, the default is to proceed. Surgical oncologists have several concerns about vaccinating their patients after major surgical procedures. Patients with cancer have impaired immunity, and the ability of our patients to mount an effective immune response to the vaccine is unclear. Conversely, due to their immunocompromised state, our patients may be more susceptible to complications from the vaccine, such as influenza-like-illness (ILI), or have higher rates of postoperative complications due to the additional immune challenge of the vaccine. Previous studies have evaluated the flu vaccine in patients receiving chemotherapy, or after organ transplantation, but the combination of cancer and major surgery remains unstudied.

This is a collaborative study with Infectious Diseases and Microbiology to evaluate the response to the flu vaccine in patients with pancreatic or gastric cancer, soft tissue sarcoma or peritoneal surface disease (i.e. carcinomatosis from appendiceal or colon cancers). Patients will be randomly selected to receive the vaccine either 2 weeks preoperatively or postoperatively at the time of discharge. Serum antibody response, rates of ILI and post-op complications will be analyzed. The long term goal of this study is two-fold: to determine the optimal time to vaccinate this group of patients in relation to their surgery, and to improve compliance with vaccination.

ELIGIBILITY:
Inclusion Criteria:Patients with gastric or pancreatic cancer, soft tissue sarcoma or peritoneal surface malignancy who will undergo surgery with curative intent are eligible.

-

Exclusion Criteria:Those with a contraindication to vaccination, patients who have a splenectomy (whether planned or not) and those who have had the flu for the year are not eligible.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-06 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Antibody Titer | Baseline
  Serum antibody titers will be assessed prior to vaccination.
Antibody Titer | 2 weeks
  Serum antibody titers will be assessed 2 weeks after vaccination
Antibody Titer | 4 weeks
  Group A will have a late titer assessed, 4 weeks after vaccination

SECONDARY OUTCOMES:
Influenza-Like-Illness | 2 weeks
  All subjects will be assessed for influenza-like-illness with a questionnaire 2 weeks after vaccination.
Surgical complications | 30 days post op
  Any postoperative complications will be recorded, specifically wound infection, pneumonia, reintubation,sepsis, MI, PE,and anastomotic leak.

CONTACTS AND LOCATIONS:
Overall Officials: Colette R Pameijer, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook Hospital, Stony Brook, New York, United States

REFERENCES:
- [Derived] Hirsch C, Zorger AM, Baumann M, Park YS, Brockelmann PJ, Mellinghoff S, Monsef I, Skoetz N, Kreuzberger N. Vaccines for preventing infections in adults with solid tumours. Cochrane Database Syst Rev. 2025 Apr 16;4(4):CD015551. doi: 10.1002/14651858.CD015551.pub2. PMID 40237463